CLINICAL TRIAL: NCT03695679
Title: Evaluation of an Interactive Web-based Sexual Health Literacy Program to Safe Sex Practice for Female University Students: A Multicentred Randomized Controlled Trial
Brief Title: Interactive Web-based Sexual Health Literacy Program and Safe Sex Practice in University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other); The Hong Kong Polytechnic University (Other); Hong Kong Shue Yan University (Other); City University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Janet Wong, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14150971
Record Dates: First submitted 2018-09-16; First posted 2018-10-04 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Safe Sex
Keywords: computer-assisted instruction/methods; safe sex; students; universities
MeSH Terms: conditions — Safe Sex

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Interactive computer-based intervention
  Interventions: Behavioral: Interactive computer-based intervention
- Control group (No Intervention): An one-page online information about procedures and tips of condom use with minimal intervention

INTERVENTIONS:
Behavioral: Interactive computer-based intervention — There are 4 components of the Interactive computer-based intervention(ICBI) which will be delivered in 3 phases:
  1. Perceived Susceptibility and Perceived Severity
  2. Perceived Benefits and Perceived Barriers
  3. Cue to Action
  4. Self-Efficacy
  In addition, a discussion forum will be created to handle questions from the participants. Also, there will be an email address for enquiries if the participants need any support or if they want to seek further enquiry/ clarification after reading the web-based information.
  Arms: Intervention group

SUMMARY:
The primary objective is to evaluate the efficacy of an Interactive web-based sexual health literacy program to enhance safe sex practice among female university students. Based on Health Belief Model, the intervention comprising: (1) personalized perceived susceptibility and perceived severity of STIs and cervical cancer; (2) perceived benefits and perceived barriers of safe sex practice via knowledge- based information; (3) cue to action via the local resources; and (4) self-efficacy via narrative stories, which are tailored for female university students, to communicate safe sex messages. The investigators hypothesised that the intervention will enhance consistency of condom use, knowledge, attitude, norms, self-efficacy towards condom use, sexual consent, sexual communication and reduce sexual coercion and casual sex among participants in intervention group compared to those in control group.

A multicentered randomized controlled trial will be conducted in 500 female university students in 5 universities with dormitories. Inclusion criteria are unmarried female university Chinese students aged at least 18-year and not received any sexual health intervention in the past 12 months. The main outcome measures will be self-reported consistency of condom use with every partner in 3-month assessments, sexual coercion, sexual consent, casual sex and sexual communication. The study instruments used will be UCLA Multidimensional Condom Attitudes Scale; Sexual Consent Scale-Revised; Conflict Tactic Scale-Revised; and Sexual Communication Self-Efficacy Scale. The data analysis will be a linear mixed effects model with intervention group and baseline consistency of condom use as the covariates. The investigators expected that the intervention will enhance consistency of condom use with Cohen effect size of 0.3.

DETAILED DESCRIPTION:
Subject recruitment procedures:

Recruitment of participants will be conducted by using bulk electronic mails, promotional brochures, posters and campus booths. An invitation card with a QR code of the web-based intervention will be used for inviting female university students to enrol the study. Online enrolment will be done for screening participants for eligibility. From the investigators' past experience in recruiting university students, the investigators shall be able to reach over 30,000 female university students in five universities.

Participants will be asked to complete the web-based baseline survey at enrolment. The web-based questionnaire will be set up under an online platform. Participants may use their mobile devices including laptop computers and smartphones to complete the questionnaire. Participation is entirely voluntary. Written informed consent will be obtained via the web-based platform before completing the baseline questionnaire.

After completion of the questionnaire, the recruited students will then be randomized to either intervention group or control group, according to a list prepared by blocked randomization of a size decided by a randomizer. The block size and order of allocation will be kept securely in the randomizer to avoid selection bias. Allocation concealment will be done at the online platform according to the participants' enrolment sequence. The participants will then be guided to a web-page according to their group allocation.

At 3-month and 6-month after the entry of the study, participants will receive a link through their e-mail to complete a follow-up questionnaire (T2). Three months later, another e-mail link will be sent to participants for completing the last follow-up questionnaire (T3). If no response from a participant, a follow-up telephone text-message and/or telephone call will be sent after 1 week as a reminder.

Sample size assessment:

Female university students (n = 500), across disciplines and year of study, will be recruited from five universities with dormitory or residential halls in Hong Kong. The sample size calculation is based on the primary comparison of behavioural change in consistency of condom use. A previous study showed the mean percentage of condom use was 67.8% (SD 39.3%) in people under an ICBI and 23.5% (SD 35.3%) in those under usual care, corresponding to a moderate to large Cohen effect size of 0.6.(20) To detect a conservative small Cohen effect size of 0.3 with 80% power and maximum 5% false positive error rate by a two-sided two-sample t-test, the investigators need a total of 352 (176 per group) female university students. Assuming 30% attrition based on a previous study using web-based intervention (21), the investigators plan to recruit a total of 500 female university students.

Quality assurance plan:

The web-based intervention is password-protected and "Pseudo-Codes" will be used to ensure anonymity and confidentiality to minimize social desirability of the responses. By asking the participant to create his/her own "pseudo-code", a code that can be accurately retyped each time the participant completes pre-test and post-test. There will otherwise no other vulnerable subjects involve in the study.

Data check and analysis method:

To assess the efficacy of ICBI in increasing consistency of condom use, a linear mixed effects model will be adopted with intervention group and baseline consistency of condom use as the covariates. The group by time interaction shall be assessed for changes of ICBI effects over time. When the interaction effect is insignificant, it will be removed from the model and the overall ICBI will be estimated. Otherwise, liner contrasts will be used to assess the ICBI effect at each time epoch. In case of baseline imbalance, additional analysis with adjustment of variables that show imbalance at baseline will be performed. If the data will not normally distributed, the corresponding analyses methods, such as zero/one inflated beta (ZOIB) regression model, will be applied based on the data characteristics.

The intention-to-treat principle will be adopted and all study subjects will be included in the analysis. Missing values at 3- and 6-month follow-up will be replaced by the last observed value and multiple imputation. Missing values at baseline will be replaced by values from 3-month or 6-month follow-up. If there will be no value obtained at any of the 3 time points, the participant will be excluded from the analysis. For other outcomes, the t test will be applied for continuous data and the chi-square test will be applied for categorical data. The analysis will be performed by using the R software (version 3.6.1; R Core Team). Each estimated effect will be accompanied by a 95% confidence interval and 5% level of significance. Questions will be downloaded from the inquiry system. Content analysis will be performed to categorise the collected responses.

Data collection and management:

The investigators and the research assistants of the research team are responsible for data collection and they will be permitted to access to source data and study record. Daily logs will be recorded by the research assistants to monitor the study progress including the number of respondents approached, interviews completed or refused and incomplete interviews. All data entered in the database will be verified and cleaned. After completion of data entry, computer logic checks will be run for consistency of related code. Necessary corrections will be made to the database.

ELIGIBILITY:
Inclusion Criteria:

* Female university students aged at least 18 years
* Able to read Chinese or understand Cantonese
* Unmarried
* Having intimate partners in the past 12 months
* Did not receive any sexual health information including formal face-to-face or online education/ training courses related to contraceptives and sexually transmitted diseases from university, hospitals, clinics and non-governmental organizations in the past 12 months

Exclusion Criteria:

* Unwilling to complete the questionnaires at 3 time points
* Pregnant women and postnatal women
* With psychiatric illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 781 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Change from consistency in condom use with every partner at 3 months | Baseline, 3-month post intervention and 6-month post intervention
  It will be assessed by using percentage of male condom protected sex with every partner according to the recommended guidelines from the systematic review of 56 studies. Other behavioural items will also be asked, for examples, condom use at last sex and description of sexual partners (dating partner vs casual partner) at last sex.

SECONDARY OUTCOMES:
Knowledge, attitude, norms and self-efficacy of condom use | Baseline, 3-month post intervention and 6-month post intervention
  It will be assessed by 25-item MCAS which contains assessment on five subscales: reliability and effectiveness of condoms, sexual pleasure associated with condom use, stigma associated with people proposing or using condoms, embarrassment about negotiating and using of condoms, and embarrassment about purchasing condoms. The measurement can be used with participants who do and do not have personal experience with condoms. The items are answered by a 7-point Likert-scale and total scores are ranged from 7 to 175. The higher the score, the more positive is the knowledge, attitude, norms, and self-efficacy of condom use.
Knowledge, attitude, norms and self-efficacy of sexual coercion and sexual consent | Baseline, 3-month post intervention and 6-month post intervention
  It will be assessed by 39-item SCS-R. It contains four attitudinal subscales (positive attitude towards establishing consent, lack of perceived behavioral control, relationship length norms, and (pro) assuming consent) and two behavioral subscales (indirect consent behaviors and awareness of consent). It is suitable for both participants who do and do not have personal experience with sexual consent. The items are answered by a 7-point Likert-scale and total scores are ranged from 39 to 273. The higher the score, the more positive is the attitude, norms, and perceived behavioural control of sexual consent.
Sexual coercion | Baseline, 3-month post intervention and 6-month post intervention
  It will be measured by 7-item subscale from Revised Conflict Tactic Scale. The responses will be on a dichotomous scale for assessing sexual coercion. All items will be rated on a 7-point Likert scale indicating how often the behaviour occurred. The higher the score, the greater the frequency.
Self-efficacy in sexual communication | Baseline, 3-month post intervention and 6-month post intervention
  It will be assessed by 20-item SCSES. It contains five domains (contraceptive communication, positive sexual messages, negative sexual messages, sexual history, and condom negotiation). The items are answered by a 4-point Likert-scale and total scores are ranged from 20 to 80. The higher the score, the more the self-efficacy in sexual communication.
Retention of the participant | 6-month post intervention
  It will be evaluated by recording retention of the participants.
Engagement time of the participants | 6-month post intervention
  It will be evaluated by recording the total time spent on the website.
Incidence of adverse events of the intervention | 6-month post intervention
  It will be evaluated by recording the adverse events of the intervention.
Overall satisfaction of the intervention | 6-month post intervention
  It will be evaluated by recording overall satisfaction of the intervention in a scale of 0-10 and overall perception of the intervention with a 5-Likert-scale. Also, participants will be asked whether they will recommend the intervention to friends and "yes" will be scored 1 point. The higher the score, the higher overall satisfaction of the intervention.
Total pages of the website each participant visited | 6-month post intervention
  It will be evaluated by recording the total pages of the website each participant visited.
Percentage of performance on the interactive tasks | 6-month post intervention
  It will be evaluated by recording each participant's performance on the interactive tasks.
Incidence of searching more information about safe sex practice | 3-month post intervention and 6-month post intervention
  Participants will be asked whether they searched for more information about safe sex practice during the last three months.
Demographics | Baseline, 3-month post intervention and 6-month post intervention
  It includes items such as gender, age, year of study, and dating relationships status. Also, the participants will be asked for history of childhood sexual coercion. The item is extracted from Adverse Childhood Experiences questionnaire - "Did an adult or person at least 5 years older than you ever touch or fondle you or have you touch their body in a sexual way? Or attempt or actually have oral, anal, or vaginal intercourse with you?" Also, the information regarding individual risks on STIs and cervical cancer will be collected at baseline (including age, age at first sexual intercourse, number of sexual partners during one's lifetime, frequency of condom use, history of ever being diagnosed with an STI, smoking status, history of giving birth, and history of having pap smear test).

CONTACTS AND LOCATIONS:
Overall Officials: Janet Yuen Ha Wong, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Nursing, LKS Faulty of Medicine, The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Zhang W, Wong CKH, Xin Y, Fong DYT, Wong JYH. A Web-Based Sexual Health Intervention to Prevent Sexually Transmitted Infections in Hong Kong: Model-Based Cost-Effectiveness Analysis. J Med Internet Res. 2023 Aug 10;25:e45054. doi: 10.2196/45054. PMID 37561571
- [Derived] Wong JY, Zhang W, Wu Y, Choi EPH, Lo HHM, Wong W, Chio JHM, Tam HLC, Ngai FW, Tarrant M, Wang MP, Ngan HY, Fong DY. An Interactive Web-Based Sexual Health Literacy Program for Safe Sex Practice for Female Chinese University Students: Multicenter Randomized Controlled Trial. J Med Internet Res. 2021 Mar 12;23(3):e22564. doi: 10.2196/22564. PMID 33709941

DOCUMENTS (1):
  • Informed Consent Form (2016-12-30): https://cdn.clinicaltrials.gov/large-docs/79/NCT03695679/ICF_000.pdf